CLINICAL TRIAL: NCT04845841
Title: Single Center, Randomized, Open-label, Cross-over Study to Investigate the Pharmacokinetics of Two Oral Formulations of Elinzanetant After Single Dosing in Healthy Participants
Brief Title: Comparison of the Extent to Which the Drug Given as Two Different Capsule Sizes Becomes Available to the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 21665; 2020-005715-49 (EudraCT Number)
Record Dates: First submitted 2021-04-07; First posted 2021-04-15 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Vasomotor Symptoms as a Sex Hormone-dependent Disorder in Women and Men
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receive study medication on time point 1 (Experimental): Participants will receive two single doses of elinzanetant in two different treatments in a randomized sequence (Treatment A, Treatment B).
  Interventions: Drug: Elinzanetant (BAY3427080) treatment A; Drug: Elinzanetant (BAY3427080) treatment B
- Participants receive study medication on time point 2 (Experimental): Participants will receive two single doses of elinzanetant in two different treatments in a randomized sequence (Treatment A, Treatment B).
  Interventions: Drug: Elinzanetant (BAY3427080) treatment A; Drug: Elinzanetant (BAY3427080) treatment B

INTERVENTIONS:
Drug: Elinzanetant (BAY3427080) treatment A — Single oral dose
Drug: Elinzanetant (BAY3427080) treatment B — Single oral dose

SUMMARY:
Researchers are looking for a new way to treat women who have symptoms by hormonal changes, like those that happen in women during menopause. These symptoms can include hot flashes, night sweats, and changes in blood pressure. These symptoms are caused by hormonal changes occurring during menopausal transition when women may have also changes in their monthly cycles. The menopausal transition most often begins between ages 45 and 55 and leads to menopause, a point in time 12 months after a woman's last period.

The study drug, elinzanetant, was designed to treat symptoms caused by hormonal changes. Before a new treatment can be approved for people to take, researchers perform clinical trials to better understand how this treatment works and to investigate safety.

The purpose of this study is to assess the blood levels of elinzanetant when given as 2 capsules of dose A (what is intended for further research and future commercialization) and also to compare the blood levels when given as 3 capsules of dose B (what was used for research up to now). Furthermore, researchers want to find out if taking of elinzanetant on two time points leads to differences in blood levels of elinzanetant.

This trial will be performed in healthy women aged 40 to 65 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 40 to 65 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, blood pressure, pulse rate, 12-lead electrocardiogram, body temperature, and laboratory tests.
* Non-smoker, at least from 3 months before the screening visit onwards
* Body weight of at least 50 kg and BMI within the range 18.0 and 30.0 kg/m*2 (inclusive) at screening.
* Female

  * Women of childbearing potential will have to use highly effective non-hormonal contraception when having sexual intercourse with a male partner from signing the informed consent form until 5 days after last dose of the study drug. Acceptable methods of contraception for this study are listed in protocol.
  * Women of non-childbearing potential are not required to use contraception. Non-childbearing potential is defined as

    * Postmenopausal state confirmed by follicle stimulating hormone (FSH) level >40 U/L, or above reference range from the local laboratory, or
    * Surgically sterilized by bilateral tubal ligation, or bilateral oophorectomy with or without hysterectomy documented by medical report verification

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Any clinically relevant abnormal findings in medical history and physical examination which in the opinion of the investigators, may put the participant at risk because of her participation in the trial or provide difficulties in interpreting the trial data.
* History or evidence of any clinically relevant cardiovascular, gastrointestinal, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other clinically relevant disease, as judged by the investigator.
* Pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study intervention will not be normal.
* Any medical disorder, condition or history of such that would impair the participant's ability to participate or complete this study in the opinion of the investigator.
* Known hypersensitivity to the study interventions (active substances, or excipients of the preparations).
* Known severe allergies e.g., allergies to more than 3 allergens, allergies affecting the lower respiratory tract - allergic asthma, allergies requiring therapy with corticosteroids, urticaria or significant non-allergic drug reactions.
* Relevant diseases within the last 4 weeks prior to the first study intervention administration.
* Febrile illness within 4 weeks before first study intervention administration.
* Regular use of medicines.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
AUC of elinzanetant | Period 1: Day 1-9, Day 11, Day 13, Day 15; Period 2: Day 1-7, Day 8 (follow up visit)
  AUC: Area under the concentration vs. time curve from zero to infinity after single (first) dose
Cmax of elinzanetant | Period 1: Day 1-9, Day 11, Day 13, Day 15; Period 2: Day 1-7, Day 8 (follow up visit)
  Cmax: Maximum observed drug concentration in measured matrix after single dose administration

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Approximately 2 to 3 months
Severity of treatment-emergent adverse events (TEAEs) | Approximately 2 to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical-Research-Services Mannheim GmbH, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.